CLINICAL TRIAL: NCT04401488
Title: Paediatric Post Pneumococcal Conjugate Vaccine Nasopharyngeal Carriage Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Solent NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RHM CHI0678
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: S. Pneumoniae; Pneumococcal Conjugate Vaccine
MeSH Terms: interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Prevenar 7 and Prevenar 13 — pneumococcal conjugate vaccines

SUMMARY:
The investigators intend to investigate the carriage of pneumococci and other respiratory microbes since the introduction of pneumococcal conjugate vaccines (Prevenar 7 and Prevenar 13). The principal aim is to gain a collection of samples that can be used to help investigate any changes that might occur in the epidemiology of microbes that are carried in the upper respiratory tract and which may cause respiratory disease, sepsis or meningitis after the introduction of Prevenar.

Nasopharyngeal and nasal swabs will be taken from up to 2,000 children aged 4 years and under in each year of the study. Swabs will be processed using traditional microbiology and molecular diagnostic techniques and isolated microbes such as S. pneumoniae further characterised using molecular methods. The investigators will also ask parents to complete a short questionnaire requesting: basic demographic data; vaccine history; recent illness; overseas travel and antibiotic usage.

The study will contribute to the success of the introduction of pneumococcal conjugate vaccines and will play a central role in maintaining confidence. The study will also help provide information for future vaccine policy as further vaccines are developed against microbes which cause respiratory disease, sepsis and meningitis.

DETAILED DESCRIPTION:
Streptococcus pneumoniae (the pneumococcus) is an important cause of pneumonia, meningitis and bacteraemia worldwide. The prevention of invasive pneumococcal disease (IPD) by immunisation has been a key public health priority. Conjugate vaccines have a good record of eradicating carriage of bacteria as well as protecting against disease because they evoke a T-cell dependent response. For this reason, they are also efficacious in children less than 2 years of age. The first pneumococcal conjugate vaccine, Prevenar 7, was licensed in the UK in 2001 and was added to the routine UK childhood immunisation schedule on 4th September 2006. Prevenar 13 replaced Prevenar 7 from 1st April 2010.

In the US Prevenar 7 was a successful intervention, resulting in decreases of childhood IPD by 69%, which was unsurprising considering that serotypes included in the vaccine (4, 6B, 9V, 14, 18C, 19F and 23F) had been reported to cause 70% of all IPD in young children. Decreases in IPD amongst the adult population were higher than predicted which is thought to have been due to herd immunity. Unfortunately this was also paralleled by an increase in disease caused by non-vaccine types or vaccine-related serotypes which had changed their protective capsule (undergone capsule switching) such as the acquisition of 19A capsular locus by a previously serotype 4 clone .

The introduction of Prevenar 7 into the UK childhood immunisation schedule led to a significant reduction in pneumococcal disease amongst children in the UK and early data after the introduction of Prevenar 13 suggests a further decline in pneumococcal carriage and disease due to the additional six serotypes contained within the vaccine. Recent studies in the UK have characterised collections of pneumococci in an attempt to better understand the clonal distribution of serotypes and sequence types. Such studies are important since pneumococci are highly transformable, with there being ample evidence of capsule switching and serotype replacement amongst pneumococci.

Although Prevenar 7 and 13 have been successful interventions in the UK and elsewhere, improved vaccines will be required to further control pneumococcal disease. Public Health England (previously Health Protection Agency) surveillance data of invasive pneumococcal disease has already indicated that serotype replacement has occurred after the implementation of Prevenar. The investigator's previous study, referred to here as the Southampton pneumococcal carriage study (Full name 'Understanding changes in the molecular epidemiology of pneumococci carried in the nasopharynx amongst children after the introduction of pneumococcal conjugate vaccines', REC No. 06/Q1704/105), also showed serotype replacement during the first three years of Prevenar 7 introduction. The serotypes seen during the investigator's SMART study (full name 'Analysis of the microbial community of the upper respiratory tract to support the development of effective vaccine policy', REC No. 11/SC/0518) similarly suggest the occurrence of serotype replacement in those who have had the Prevenar vaccine due to the low level of vaccine types found within the investigator's data set (data not yet published). There is currently insufficient evidence for the wider use of Prevenar 13 in teenagers and younger adults.

The introduction of vaccines that contain only selected serotypes, as is the case with Prevenar 7 and Prevenar 13, have been shown to promote S. pneumoniae capsule switching or capsule replacement which allows for the evasion of vaccine induced host immunity. It is therefore important to monitor which serotypes of S. pneumoniae are commonly causing disease. It is also important to analyse the nasopharynx as an ecological niche because a reduction in the carriage of pneumococci, due to Prevenar, could lead to a replacement effect such that pneumococci of serotypes not covered by the vaccine or other bacterial/microbe species may fill the niche. It is therefore also important to gain information on the carriage of other bacteria/microbes such as Haemophilus influenzae, Staphylococcus aureus and Neisseria meningitidis.

Many studies have been largely limited to studying disease-causing pneumococci and needed to be supplemented by pneumococcal carriage studies such as the investigator's Southampton pneumococcal carriage study. The Southampton pneumococcal carriage study started immediately before the implementation of pneumococcal conjugate vaccines in the UK and completed its eighth swabbing time-point during winter 2013/14. It was the only longitudinal pneumococcal carriage study of its kind in the UK and is, to the investigators knowledge, one of only two longitudinal carriage studies globally that began as Prevenar was being introduced, the other being in Massachusetts, USA. The investigator's SMART study gives a unique snapshot of bacterial carriage in the community in all age groups and has provided information which will enable us to better understand bacterial carriage. The investigators believe that such studies are of high importance in understanding the carriage of microbes, in particular pneumococcal carriage, during the implementation of pneumococcal conjugate vaccines.

The paediatric post pneumococcal conjugate vaccine nasopharyngeal carriage study is a development of the Southampton pneumococcal carriage study which proposes to continue to contribute to the success of the introduction of pneumococcal conjugate vaccines and, depending on the biological consequences of on-going vaccine use, play a central role in maintaining confidence. The study will also help provide information for future vaccine policy and vaccine development as further pneumococcal conjugate vaccines, and indeed other vaccines such as the meningococcal B vaccine, are introduced. Although Prevenar vaccines have been successful interventions, reducing pneumococcal deaths for children under 5 years of age globally by an estimated 250,000 between 2000 and 2008, there were still a reported 485,000 pneumococcal deaths in children of this age range in 2008 alone. Conjugate vaccines will need to be continuously redesigned in order to maintain suppression of pneumococcal disease. It is therefore important to continue gaining information on circulating serotypes and sequence types from carriage and compare these to disease-causing pneumococci since the implementation of Prevenar and relate this to the potential development and introduction of new vaccines.

Hypothesis The circulating pneumococcal population of the nasopharynx has implications for pneumococcal disease in children.

Aims

* to gain a collection of pneumococci and other microbes of related importance that can be used to help investigate any changes that occur in the epidemiology of pneumococcal disease since the introduction of Prevenar 13.
* to use microbes isolated from the respiratory tract during the investigator's previous studies (the Southampton pneumococcal carriage study and the SMART study) to further investigate the carriage of microbes including S. pneumoniae and the effects of Prevenar.
* to use all isolated strains to help understand changes in the molecular epidemiology of pneumococci, and other relevant microbe species of the upper respiratory tract.

Research questions

This study aims to provide key data that will continue to support the implementation of pneumococcal vaccines. The key outcomes from this study are:

* To contribute to understanding any changes that may take place in the frequency of nasopharyngeal carriage of the pneumococcus and microbes of related importance and, at a molecular level, how these changes may have occurred.
* To continue providing data on the molecular epidemiology of carried pneumococci in young children.
* To describe the indirect impact of Prevenar 13 on pneumococcal carriage in young children.
* To compare the genomic epidemiology of serotype 3 pneumococci in carriage and disease with the aim of identifying reasons for the ineffectiveness of Prevenar-13 against this serotype.
* To compare the genomic epidemiology of non-Prevenar 13 serotypes from carriage and disease with Prevenar 13 serotypes with the aim of identifying differences in their virulence potential.

Methods Recruitment for the paediatric post pneumococcal conjugate vaccine nasopharyngeal carriage study will take place year-round. The investigators aim to recruit children aged 4 years and under who are visiting either the Paediatric Outpatients department at University Hospital Southampton NHS Foundation Trust or Solent NHS Trust sites and sites working in partnership with the Solent NHS Trust. By analysing pneumococci and other microbes of importance collected from the Southampton pneumococcal carriage study, the SMART study and the paediatric post pneumococcal conjugate vaccine nasopharyngeal carriage study, it will be possible to examine the impact of immunisation on the pneumococcal population and overall carriage of microbes of interest in an age group at high risk of acquisition and carriage. Swabs and/or swab contents from participants and the microbes isolated from swabs from the above studies will be stored for the duration on this project. The current study is cross-sectional in order to gain a 'snapshot' of the frequency and types of pneumococci and other microbes of importance being carried amongst young children.

During the paediatric post pneumococcal conjugate vaccine nasopharyngeal carriage study, swabs from the back of the nose (Nasopharyngeal swabs) will be taken from up to 2,000 children aged 4 years and under in each year of the study. The investigators will also ask to take nasal swabs, but these will be optional. Swabs will be taken from children who are already attending/visiting the Paediatric Outpatients department at University Hospital Southampton NHS Foundation Trust or Solent NHS Trust sites and sites working in partnership with the Solent NHS Trust. Swabbing will be performed following a modified World Health Organisation (WHO) protocol. Swabs will be collected by either a trained healthcare professional (i.e. a research nurse, health care assistant, medical student, doctor) or a trained member of the study team (i.e. clinical trials assistants) and submitted to the project research team for selective bacterial isolation and testing such as molecular analysis. As was the practice for the Southampton pneumococcal carriage study and the SMART study, swabs will be taken solely for research purposes and will be anonymised immediately; there will be no patient identifier on the swabs. Swabs will be taken to the research team at University Hospital Southampton NHS Foundation Trust and processed within 48 hours of being taken. The remaining contents of new swabs collected as part of the study will be stored in microbial storage media for the future analysis of microbe DNA only - no human DNA will be analysed at any time. At this stage the swabs will be disposed of using the normal practices of University Hospital Southampton NHS Foundation Trust. The selective media plates will be examined after incubation for the presence of Streptococcus pneumoniae, Staphylococcus aureus, Haemophilus influenzae, α haemolytic Streptococcus, Neisseria meningitidis and Moraxella catarrhalis. If a plate shows growth of any of these bacteria, individual colonies will be sub-cultured and subsequently frozen for future analysis e.g. to determine the frequency of carriage of multiple serotypes and sequence types. Any bacteria/microbes isolated will be deemed a gift to the research study. This information is given on the patient information sheet. If a participant withdraws from the study the bacteria isolated from their swab will be destroyed.

The investigators will also ask parents/ guardians to complete a short questionnaire requesting basic demographic data, vaccine history, information regarding recent illness and recent antibiotic usage. This is to help allow us to understand the impact of age, demographic data and/or vaccine and antibiotic history on the carriage of specific respiratory microbes.

Analysis will be done using the bacteria isolated and swab contents stored in microbial storage media as part of this paediatric post pneumococcal conjugate vaccine nasopharyngeal carriage study, as well as bacteria isolated and stored during the Southampton pneumococcal carriage study and the SMART study to investigate carriage of microbes including S. pneumoniae and the effects of Prevenar.

Sampling and statistical power The study design is cross-sectional. Children aged 4 years and under will be sampled. Up to 1,000 participants will be recruited each winter (October to March), until winter 2019/2020, at which point year-round recruitment will be undertaken and up to 2000 participants will be recruited each year. The parents of potential participants will be approached by a trained healthcare professional or member of the study team in the reception/waiting room of the Paediatric Outpatients Department of University Hospital Southampton NHS Foundation Trust or Solent NHS Trust sites and sites working in partnership with the Solent NHS Trust. All participants will be aged 4 years and under; therefore, the parents or legal guardian will be asked to provide informed consent for their child's participation in the study. Informed consent will be taken after having time to read the information sheet provided and will therefore be based on information provided in in the information sheet and the opportunity to question study personnel. Entry to the study will be voluntary.

The investigator's previous pneumococcal carriage studies have found an average carriage rate of approximately 30%. The investigators had previously assumed that the introduction of pneumococcal conjugate vaccines would lead to a reduction in the pneumococcal carriage rate due to a reduction in serotypes included in the vaccines. Although there was a reduction in these serotypes, a concomitant increase of non-vaccine serotypes occurred. For the present study, the investigators have therefore assumed that the overall pneumococcal carriage rate will remain at 30%. In order to detect a carriage rate of 30% (with 95% CI width of 5% on both side of the carriage rate) the investigators will require at least 340 participants per winter (allowing an error rate of 5% to occur during culturing). To detect rare serotypes with a carriage rate as low as 2% (with 95% CI width of 1% on both side of the carriage rate) the investigators will require at least 793 participants per winter allowing an error rate of 5% to occur during culturing). However, since this is a pragmatic study whereby the future epidemiology of pneumococcal carriage is unknown, with or without further novel vaccine implementation, the investigators anticipate that up to 1,000 participants per winter will be required to detect significant changes the pre-specified precision in the overall pneumococcal carriage rate and/or specific serotype carriage rate. This will then enable us to detect an overall carriage rate as low as 3% (with 95% CI width of 1% on both side of the carriage rate). Increased recruitment of 2000 participants per year allows for the detection of carriage prevalence of 30% (with 95% CI width of 2% on both side of the carriage rate allowing an error rate of 5% to occur during culturing).

A power calculation was performed by a statistician at the University of Southampton.

Timetable The study started on the 10th November 2014 and will recruit/swab for 8 years (as a result of an extension given REC approval 22nd March 2016 and an extension given REC approval 2nd September 2019 and HRA approval 23rd August 2019). Recruitment and swabbing took place during the winters (October to March) of 2014/15, 2015/16, 2016/17, 2017/18, 2018/19 and then year-round from October 2019 to March 2022 (as per the amendment submitted March 2020). This extended recruitment allows the year-round surveillance of S. pneumoniae to detect fluctuation of carriage. In response to the COVID-19 outbreak, it also allows the detection of circulating microbes of outbreak, epidemic and pandemic potential. The study will end 31st March 2027 to allow enough time for analysis.

All sampling will take place within the Outpatients Department of University Hospital Southampton Foundation NHS Trust (or the NIHR Clinical Research Facility if there are no rooms available in the Outpatients Department) or at Solent NHS Trust sites and sites working in partnership with the Solent NHS Trust. Academic work will take place within the Faculty of Medicine, University of Southampton and at collaborating centres such as the Wellcome Trust Sanger Institute, Cambridge.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 4 years or under, attending the recruitment sites during the recruitment period will be invited to participate through their parents or legal guardian.

Exclusion Criteria:

* One child per family
* Children with obstructed nasal passages

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 4 years and under.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Collection of pneumococci | By the end of the study (31/03/2027)
  To gain a collection of pneumococci and other microbes of related importance that can be used to help investigate any changes that occur in the epidemiology of pneumococcal disease since the introduction of Prevenar 13

SECONDARY OUTCOMES:
Understand changes in the molecular epidemiology of pneumococci | By the end of the study (31/03/2027)
  To use all isolated strains to help understand changes in the molecular epidemiology of pneumococci, and other relevant microbe species of the upper respiratory tract.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton Foundation NHS Trust, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No